CLINICAL TRIAL: NCT04576624
Title: A Brain-Health Lifestyle Restructuring Intervention for Older Adults With Mild Cognitive Decline : Feasibility, Effectiveness, and Experiences With the Intervention
Brief Title: Brain-Health Lifestyle Restructuring Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng Kung University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Ling-Hui Chang, Associate Professor, National Cheng Kung University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: National Cheng-Kung University
Record Dates: First submitted 2020-09-08; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Lifestyle; Cognitive Decline; Aging
Keywords: lifestyle intervention; brain health; aging; cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: three-year project using a combined pragmatic randomized controlled clinical trial and multiple case studies mixed-method research design
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lifestyle Intervention (Experimental): Subjects in the Lifestyle Intervention group will, in six months, receive sixteen group sessions and six individualized treatment sessions.
  Interventions: Behavioral: Lifestyle Intervention
- Social Activities (Sham Comparator): Social Activities Group will receive twenty-two group sessions
  Interventions: Behavioral: social activity
- Passive Control (No Intervention): Control group will receive patient education materials with each assessment

INTERVENTIONS:
Behavioral: Lifestyle Intervention — A combined approach of a lifestyle structuring intervention to improve the general health and quality of life of persons with cognitive impairments. The investigators propose to combine a multi-modal cognitive intervention and lifestyle redesign approach to improve the cognitive health of older persons with cognitive impairments.
  Arms: Lifestyle Intervention
Behavioral: social activity — 24 social gathering events
  Arms: Social Activities

SUMMARY:
With population aging, the number of older persons with cognitive impairments increases. Literature support the effectiveness of a lifestyle approach to promote the health of persons with cognitive impairment, as well as a Lifestyle Redesign intervention to improve the general health and quality of life of frail older adults. The investigators propose to combine a multi-modal cognitive intervention and lifestyle redesign approach to improve the cognitive health of older persons with cognitive impairments.

DETAILED DESCRIPTION:
With population aging, the number of older persons in Taiwan with cognitive impairments increases. Recent years witnessed an expansion of governmental policies and services dedicated to improve long-term care. It is critical to develop an effective cognitive intervention that can prevent, delay, or slow down cognitive decline. Although literature support a multi-modal approach to preserve the cognitive capacity of older adults with cognitive impairments, there is inadequate attention to facilitate the integration of cognitively therapeutic activities to daily routines, nor to the establishment of a lifestyle that promote brain health. Therefore, the adherence to the intervention program was low after the program ended.

Literature support the effectiveness of a lifestyle approach to promote the health of and reduce medical cost for persons with chronic diseases, such as cardiovascular diseases and diabetes. Empirical evidence also supports the effectiveness of Lifestyle Redesign intervention to improve the general health and quality of life of frail older adults. The investigators propose to combine a multi-modal cognitive intervention and lifestyle redesign approach to improve the brain health of older persons with cognitive impairments. The goals of this project are thus three-folds:

1. To develop a contextualized lifestyle restructuring intervention that facilitates the integration of cognition-promoting activities into daily routines and examine the feasibility of this intervention.
2. To compare the effectiveness of a brain-health lifestyle restructuring intervention, social activity, and passive control in (1) general cognition, activity participation, activities of daily living function, and quality of life, and (2)physical function and cognitive function at the end of the intervention, 6 months after, and one year after.
3. To qualitatively explore the experiences of the participants with the intervention, perceived effectiveness, and its contextual influences.

This is a three-year project using a combined pragmatic randomized controlled clinical trial and multiple case studies mixed-method research design. One hundred twenty-two older adults with cognitive impairments and residing in community will be recruited and randomly assigned to the groups of Lifestyle Intervention, Social Activities, and Passive Control. Subjects in the Lifestyle Intervention group will, in six months, receive sixteen group sessions and six individualized treatment sessions. Social Activities Group will receive twenty-two group sessions. Control group will receive patient education materials with each assessment. All participants will receive pre- and post-intervention, 6-month, and 12-month follow-up evaluations. Primary outcomes include cognitive function, activity participation, daily activity functions , and quality of life. Secondary outcomes include physical function, functional memory, working memory, complex attention, and processing speed.

Descriptive statistics, inferential statistics, factorial ANNOVA, and Generalized Estimating Equation will be used to evaluate and compare the effectiveness of the Lifestyle Restructuring Intervention. This study will also use multiple case studies to qualitatively understand the experiences of eight participants about their participation in the intervention, cognitive decline, and the contextual factors that affects their participation. Sequential interviews and participant observation will be used to do qualitative data collection.

ELIGIBILITY:
Inclusion Criteria:

* Over 55 years old and living in the community
* Reported cognitive declines.

Exclusion Criteria:

* Within normal cognition, determined by scoring more than 24 in the Taiwanese version of the Montreal Cognitive Assessment
* Having any medical, neurological, psychiatric conditions, and depression by scoring above 10 in the Brief Symptom Rating Scale
* Having severe visual, auditory, speech or physical problems that limit them to follow instructions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | pre-intervention
  Montreal Cognitive Assessment, with a value of 0-30. Higher scores mean a better outcome.
Cognitive function | 6 months after the intervention begins
  Montreal Cognitive Assessment, with a value of 0-30. Higher scores mean a better outcome.
Cognitive function | 6 month after the end of intervention
  Montreal Cognitive Assessment, with a value of 0-30. Higher scores mean a better outcome.
Activity participation | pre-intervention
  Canadian Performance of Occupational Performance, with a value of 0-10. Higher scores mean a better outcome.
Activity participation | 6 months after the intervention begins
  Canadian Performance of Occupational Performance, with a value of 0-10. Higher scores mean a better outcome.
Change of activity participation | 6 month after the end of intervention
  Canadian Performance of Occupational Performance, with a value of 0-10. Higher scores mean a better outcome.
QOL (Quality of Life) | pre-intervention
  COOP/WONCA is the full title of the assessment. The assessment has a value of 6-30. Higher scores mean a poorer outcome.
QOL (Quality of Life) | 6 months after the intervention begins
  COOP/WONCA is the full title of the assessment. The assessment has a value of 6-30. Higher scores mean a poorer outcome.
QOL (Quality of Life) | 6 month after the end of intervention
  COOP/WONCA is the full title of the assessment. The assessment has a value of 6-30. Higher scores mean a poorer outcome.

SECONDARY OUTCOMES:
Physical function | pre-intervention
  Short Physical Performance Battery
Physical function | 6 months after the intervention begins
  Short Physical Performance Battery has a scale of 0-12, higher score indicating a better outcome.
Physical function | 6 month after the end of intervention
  Short Physical Performance Battery has a scale of 0-12, higher score indicating a better outcome.
Functional memory | pre-intervention
  Contextual Memory Test with a score of 0-20, with higher score indicating a better outcome.
Functional memory | 6 months after the intervention begins
  Contextual Memory Test with a score of 0-20, with higher score indicating a better outcome.
Functional memory | 6 months after the end of intervention
  Contextual Memory Test with a score of 0-20, with higher score indicating a better outcome.
Working memory | pre-intervention
  Digit Forward and Digit Backward with a score of 2-10, , with higher score indicating a better outcome.
Working memory | 6 months after the intervention begins
  Digit Forward and Digit Backward with a score of 2-10, , with higher score indicating a better outcome.
Working memory | 6 months after the end of intervention
  Digit Forward and Digit Backward with a score of 2-10, , with higher score indicating a better outcome.
Complex attention | pre-intervention
  The score of Color Trail Test-1 & 2 is the time spent to complete the test. The test will be terminated when 4 minute is up. Lesser time indicates a better outcome.
Complex attention | 6 months after the intervention begins
  The score of Color Trail Test-1 & 2 is the time spent to complete the test. The test will be terminated when 4 minute is up. Lesser time indicates a better outcome.
Complex attention | 6 months after the end of intervention
  The score of Color Trail Test-1 & 2 is the time spent to complete the test. The test will be terminated when 4 minute is up. Lesser time indicates a better outcome.
Processing speed | pre-intervention
  Symbol Digit Substitution Test takes 90 seconds to complete. The score is the number of correct responses. A higher score indicates a better outcome.
Processing speed | 6 months after the intervention begins
  Symbol Digit Substitution Test takes 90 seconds to complete. The score is the number of correct responses. A higher score indicates a better outcome.
Processing speed | 6 months after the end of intervention
  Symbol Digit Substitution Test takes 90 seconds to complete. The score is the number of correct responses. A higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Hui Chang, Principal Investigator — Department of Occupational Therapy, NCKU
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No